CLINICAL TRIAL: NCT01323504
Title: Pain and Music Therapy During the Wound Healing in Patient Suffering Arteritis of Stage 5 or 6.
Brief Title: Pain and Music Therapy in Patients Suffering Arteritis
Acronym: Musicthérapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Marc LASKAR, CHU de Limoges
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: I09022 / musicthérapy
Record Dates: First submitted 2011-03-15; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Arteritis
Keywords: Stage 5 arteritis; Stage 6 arteritis; rutherford classification
MeSH Terms: conditions — Arteritis | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy group (Experimental): Local care with music
  Interventions: Other: Music
- control group (No Intervention): Local care without music
  Interventions: Other: no music

INTERVENTIONS:
Other: Music — Patient are listen music during their local care
  Arms: Music therapy group
Other: no music — There are no music during the local care
  Arms: control group

SUMMARY:
It is estimated that 800,000 people in France suffer from peripheral artery disease (PAD), of whom 1-2% present the most severe form critical limb ischaemia (CLI). In this situation, the patient frequently presents painful non-healing ulcers and focal gangrene. Wound care is generally associated with increasing pain. Pain relief may be challenging in spite of major analgesics.

Several studies in this country and elsewhere assessed the usefulness of music for chronic or acute pain relief during care. However, no data are published regarding the interest of music therapy for pain relief during local care in PAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged at least 18 years, affiliated to the health insurance scheme.
* Patients affected by arteritis of stage 5 or 6 at Limoges University Hospital in department cardiovascular Surgery.
* Patients requiring a daily repair of bandage, not exceeding fifteen minutes and provoking a pain
* Initial pain equal to three during local care in the digital scale.
* Having given their enlightened consent writes

Exclusion Criteria:

* Bypass and / or angioplasty lower than one week
* Diabetic neuropathy
* Patient who is going to undergo a surgery of amputation
* Patients affected by demented pathologies or by confusion
* Pregnant or breast-feeding women or without effective contraception
* Patients being the object of a saving of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief during local care with music or not. | 7 days
  Different level of pain front-counterpart realization of the bandage which will be compared between both groups of patients in the seventh day after implementation of the procedure. The level of pain will be measured by a digital scale from 0 to 10.

SECONDARY OUTCOMES:
Quantification in equivalent morphine of the analgesic prescription at the seventh day | 7 days
  * Quantification in equivalent morphine of the analgesic prescription at the seventh day after implementation of the musicotherapy
  * Pain intensity during the bandage at the seventh day measured by digital scale from 0 to 10.
  * anxiety intensity at the seventh day measured by scale HAD after implementation of the musicotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Marc LASKAR, MD, Principal Investigator — University Hospital, Limoges